CLINICAL TRIAL: NCT01204320
Title: A COMparison Between PAClitaxel-coated Balloon and pacliTaxel-eluting Stent in the Treatment of In-Stent Restenosis (COMPACT-ISR)
Acronym: COMPACT-ISR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale San Donato (Other)
Responsible Party: Cardiovascular Department USL 8(Leonardo Bolognese MD), Ospedale SanDonato
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Arezzo003
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2009-10

CONDITIONS: Stable Angina; Unstable Angina
Keywords: Restenosis; POBA; Stenting; Paclitaxel
MeSH Terms: conditions — Angina, Stable; Angina, Unstable

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel-coated Balloon (Experimental): Paclitaxel-coated Balloon Angioplasty
  Interventions: Procedure: Paclitaxel-coated Balloon
- Paclitaxel-eluting Stent (Active Comparator): Paclitaxel-eluting Stent Implantation
  Interventions: Device: Paclitaxel-eluting Stent

INTERVENTIONS:
Procedure: Paclitaxel-coated Balloon — POBA
  Other Names: Orbus
  Arms: Paclitaxel-coated Balloon
Device: Paclitaxel-eluting Stent — Stenting
  Other Names: Taxus
  Arms: Paclitaxel-eluting Stent

SUMMARY:
This is a multicentric randomized comparison between paclitaxel-coated balloon angioplasty or paclitaxel-eluting stent implantation in patients with stable or unstable angina with the evaluation of restenosis by Quantitative Coronary Analysis.

DETAILED DESCRIPTION:
The purpose of this study is to determine the late luminal loss by Quantitative Coronary Analysis at 6 month-follow up after paclitaxel-coated balloon angioplasty or paclitaxel-eluting stent implantation in the treatment of in-stent restenosis.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* >18y
* Stable Angina or Unstable Angina
* Single restenotic lesion in a previously stented coronary artery

Exclusion Criteria:

* Acute Myocardial Infarction within 72h
* Serum Creatinine>2.0 mg/dL
* Contraindications to ASA, Heparin, Clopidogrel, Ticlopidine, Abciximab, Tirofiban, Paclitaxel
* Contraindications to contrast media
* Life expectancy < 2y
* Target Lesion length > 30mm
* Target Lesion diameter <= 2.5 mm
* Target stenosis < 70%
* Massive Calcifications in the target segment
* Evidence of intra-coronary thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Late Luminal Loss defined as the difference between the minimal luminal diameter after stenting and at follow-up by Quantitative Coronary Analysis | 6 months

SECONDARY OUTCOMES:
Binary restenosis defined as >50% diameter stenosis by QCA | 6 months
Major Adverse Cardiac Events | 6, 12 months
Target Lesion Revascularization | 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Bolognese, MD, Study Chair — Cardiovascular Department - San Donato Hospital
Locations (1):
- San Donato Hospital, Arezzo, AR, Italy